CLINICAL TRIAL: NCT03720288
Title: Prospective Analysis Between Acetazolamide vs Placebo in Patients With Acute Heart Failure
Brief Title: Acetazolamide in Patients With Acute Heart Failure
Acronym: ACETA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSInCor-Acetazolamide
Record Dates: First submitted 2018-10-19; First posted 2018-10-25 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure; Acute Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetazolamide (Experimental): All patients will receive an initial dose of intravenous furosemide of 1mg / kg, subsequently descaled to 0.5mg / kg of 6 / 6h, associated with oral hydrochlorothiazide 25mg / day and spironolactone 25mg / day orally. When the patient is randomized to the acetazolamide group, he / she will start using the adjuvant medication as acetazolamide drug capsule at the daily dose of 250 mg / day (oral) during the first three days of treatment.
  Interventions: Drug: Acetazolamide
- Placebo (Experimental): All patients will receive an initial dose of intravenous furosemide of 1mg / kg, subsequently descaled to 0.5mg / kg of 6 / 6h, associated with oral hydrochlorothiazide 25mg / day and spironolactone 25mg / day orally. When the patient is randomized to the placebo group, he / she will start using the placebo drug capsule during the first three days of treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — Patient will follow the treatment according to inclusion sequence, receiving the corresponding number medication.
  Arms: Acetazolamide
Drug: Placebo — Patient will follow the treatment according to inclusion sequence, receiving the corresponding number medication.
  Arms: Placebo

SUMMARY:
Introduction: Recent studies have suggested that the use of acetazolamide may assist in the vol- ume management of patients with decompensated heart failure (HF). However, prospective and randomized comparison in patients with HF and optimized diuretic therapy has not been described. Objective: The aim of this study was to evaluate the effectiveness and safety of the use of acetazolamide versus placebo in volume control in patients with decompensated HF. Methodology: For this, a unicentric, randomized, double blind and prospective study will be performed in a comparative manner. Hospital data (test results, medical outcomes, drug dose, complications) of patients will be analyzed for safety and effectiveness. Expected results: The use of acetazolamide as an adjuvant treatment is superior to the standard strategy for volume control in patients with decompensated HF.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women aged> 18 years.
* Patients with LVEF ≤ 40% documented on echocardiography
* BNP> 500 pg / mL
* Signed consent form.

Exclusion Criteria:

* Pregnancy
* COPD
* Hepatical cirrhosis
* Known allergy to acetazolamide
* 2nd or 3rd degree atrioventricular block.
* SBP <90 mmHg or need for vasopressor / inotropic use.
* Body mass index greater than 40 kg / m2.
* Acute coronary syndrome.
* Orotracheal intubation.
* Presence of significant pericardial effusion.
* Left ventricular outflow tract obstruction.
* Serum creatinine> 5.0 mg / dL, creatinine clearance <10 mL / min or hemodialysis.
* Presence of 2 or more clinical / laboratory / radiological criteria of infection defined by:

  * Fever
  * Leukocyte> 12,000 / mm3 or> 10% of young forms,
  * Disuria
  * Productive cough
  * Bacteremia
  * Inflammatory / infectious skin lesions
  * Abdominal pain with signs of peritonitis
  * Radiological image of pneumonia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
diuresis and negative water balance | 72 hours
  The comparison between groups for diuresis and negative water balance

SECONDARY OUTCOMES:
Number of cases with worsening of renal function | 72 hours
  worsening of renal function (increase of 0.5 mg / dl or 25% increase in relation to admission creatinine)
Number of cases with lowering of consciousness level | 72 hours
  lowering of consciousness level
Number of cases with circulatory assistance | 72 hours
  need for mechanical circulatory assistance
Number of cases with vasopressor | 72 hours
  need for vasopressor or inotropic association
Number of cases with orotracheal intubation | 72 hours
  need for orotracheal intubation
Number of cases with arrhythmia | 72 hours
  occurrence of sustained ventricular arrhythmia
Number of cases with acetazolamide side effects | 72 hours
  need for suspension of acetazolamide due to side effects
Number of cases of death | 72 hours
  ocurrence of death
Level of Base excess | 30 days
  Comparison of all hemodynamic / metabolic parameters to be evaluated (base excess)
Level of bicarbonate | 30 days
  Comparison of all hemodynamic / metabolic parameters to be evaluated
Rate of systolic and diastolic blood pressure | 30 days
  Comparison of all hemodynamic / metabolic parameters to be evaluated
Level of cardiac output | 30 days
  Comparison of all hemodynamic / metabolic parameters to be evaluated
Level of systolic volume | 30 days
  Comparison of all hemodynamic / metabolic parameters to be evaluated
Level of arterial lactate | 30 days
  Comparison of all hemodynamic / metabolic parameters to be evaluated
Level of BNP | 30 days
  Comparison of all hemodynamic / metabolic parameters to be evaluated
Level of troponin | 30 days
  Comparison of all hemodynamic / metabolic parameters to be evaluated
heart rate | 30 days
  Comparison of all hemodynamic / metabolic parameters to be evaluated
Level of sodium | 30 days
  Comparison of all hemodynamic / metabolic parameters to be evaluated
Level of potassium | 30 days
  Comparison of all hemodynamic / metabolic parameters to be evaluated
Level of creatinine | 30 days
  Comparison of all hemodynamic / metabolic parameters to be evaluated
Level of urea | 30 days
  Comparison of all hemodynamic / metabolic parameters to be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Mucio Tavares, MD, Principal Investigator — Unidade Clínica de Emergência
Locations (1):
- Instituto do Coração - HMFMUSP, São Paulo, Brazil